CLINICAL TRIAL: NCT03839550
Title: The Multi-center, Randomized and Controlled Phase II Trail of Apatinib Mesylate Tablets Combined With PD-1 Antibody SHR-1210 for Adjuvant Treatment of Patients With High Recurrence Risk After Radical Operation of Hepatocellular Carcinoma
Brief Title: Combine Apatinib Mesylate With PD-1 Antibody SHR-1210 for HCC With High Risk of Recurrence After Radical Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hong Zhao, chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAMS-HCC-SHR1210
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib Mesylate +SHR-1210 (Experimental): Experimental arm: Apatinib mesylate +PD-1 antibody SHR-1210 for adjuvant therapy of HCC with high incidence of tumor recurrence after hepatic resection
  Interventions: Combination Product: Apatinib Mesylate +SHR-1210
- Hepatic Arterial Infusion(HAI) (Active Comparator): Active Comparator arm: HAI for adjuvant therapy of HCC with high incidence of tumor recurrence after hepatic resection
  Interventions: Procedure: Hepatic Arterial Infusion(HAI)

INTERVENTIONS:
Combination Product: Apatinib Mesylate +SHR-1210 — Apatinib mesylate tablets: 250 mg, orally once a day. Take about half an hour after a meal with warm water (the daily dose should be as much as possible.
  SHR-1210: 200mg, intravenous infusion for 30 minutes (including the time of the tube, the overall infusion time is not shorter than 20 minutes, no longer than 60 minutes), once every 2 weeks. A total of 6 months of treatment,starting 4-8 weeks after radical hepatic resection.
  Arms: Apatinib Mesylate +SHR-1210
Procedure: Hepatic Arterial Infusion(HAI) — Twice standard HAI treatment, the first treatment was performed 4-8 weeks after radical hepatic resection, and the second treatment was given 4-8 weeks after the first treatment (the specific time interval depends on the recovery of liver function of the patient). The specific dosage regimen is 80-100 mg of epirubicin or 50 mg of epirubicin + oxaliplatin 50 mg per HAI treatment.
  Arms: Hepatic Arterial Infusion(HAI)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Apatinib Mesylate combined with PD-1 antibody SHR-1210 in HCC patients with high risk of disease recurrence contained microsatellite lesions, microvascular invasion(MVI) or secondary and above portal vein tumor thrombosis (PVTT) after radical resection. Patients will be randomized 1:1 either to the experimental arm to receive Apatinib Mesylate and PD-1 antibody SHR-1210 or to the standard therapy arm of hepatic arterial infusion(HAI) .

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common malignancy worldwide, which is the third cause of cancer related deaths. Radical hepatic resection is one of the most potentially curative treatments for HCC. Unfortunately, the long-term survival after radical hepatic resection is unsatisfactory because of the high incidence of tumor recurrence with the recurrence rates at 2 and 5 years are approximately 50 % to 60 % and 80 %,respectively. Microsatellite lesions, microvascular invasion (MVI) , or portal vein tumor thrombosis (PVTT) are the main risk factors for poor prognosis in HCC.

HCC is a typical vascular-rich tumor, and its occurrence, development, metastasis and invasion are closely related to angiogenesis. Due to the long-term chronic inflammatory response of the liver, the establishment and development of HCC can be induced by creating an immunosuppressive microenvironment, including up-regulation of PD-1 receptors. Therefore, immunotherapy is also considered to be a potential effective method for advanced HCC treatment. And there is little convincing evidence indicating that adjuvant therapy reduces the risk of recurrence after hepatic resection. Furthermore, no standard regimen has been established.

In the present study, we assessed the efficacy and safety of Apatinib Mesylate that is Small molecule anti-angiogenic targeted drugs /PD-1 antibody SHR-1210 combination therapy for surgically resected HCCs with high incidence of tumor recurrence containing microsatellite lesions, microvascular invasion(MVI) or secondary and above portal vein tumor thrombosis (PVTT).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old.
2. Patients were primary Hepatocellular carcinoma according to standardization of diagnosis and treatment for Hepatocellular carcinoma(2017 edition)
3. The imaging examination confirmed complete response (CR) after 1 month radical surgery ,and consented to postoperative adjuvant therapy
4. Preoperative imaging (CT/MRI/PET-CT), intraoperative or postoperative pathology confirmed HCC patients with high risk of disease recurrence contained microsatellite lesions, microvascular invation(MVI) or secondary and above portal vein branches tumor thrombosis (PVTT) after radical resection.
5. Preoperative imaging and perioperative outcomes confirmed no lymph node metastasis and distant metastasis.
6. Child-Pugh A.
7. No anti-tumor treatment before radical hepatic resection.
8. BCLC A-B
9. Eastern Cooperative Oncology Group(ECOG) body condition score 0-1.
10. Adequate main organ function:

    Hemoglobin ≥ 90g/L. Absolute neutrophil count (ANC) ≥ 1,500/mm3. Platelets ≥ 100,000/ul. Albumin ≥ 29g/L. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 the upper limit of normal (ULN). Total bilirubin (TBIL) ≤ 1.5 ULN. Creatinine ≤ 1.5 ULN.
11. Women of childbearing age (generally 15-49 years of age) are required to have a negative pregnancy test (serum or urine) within 14 days prior to enrollment, and will voluntarily use the appropriate method of contraception during the observation period and within 8 weeks after the last administration of the study drug; For men, appropriate methods of contraception should be used during the observation period and within 8 weeks after the last administration of the study drug.
12. Be willing and able to provide written informed consent for the study.

Exclusion Criteria:

1. History of liver transplantation.
2. Tumor rupture or invasion of adjacent organs.
3. History of immunosuppressive drugs used for 14 days prior to the first use of SHR-1210, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones .
4. Subjects are allergic to Apatinib Mesylate Tablets, SHR-1210, pharmaceutical excipients, o other monoclonal antibodies.
5. Attenuated Live Vaccine in four weeks before study or during study.
6. Uncontrolled or symptomatic active central nervous system (CNS) metastases (if these patients have been treated to clinically stable and discontinuation of anticonvulsants and steroids in four weeks before study may be enrolled).
7. Peripheral neuropathy grade> 1.
8. History of autoimmune disease(Subjects with vitiligo or asthma in childhood but complete remission after adult intervention after adulthood may be enrolled)
9. Subjectes diagnosed any other malignant tumor within 3 years prior to study, except for adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ
10. History of Human Immunodeficiency Virus (HIV).
11. Cardiovascular disease: Myocardial infarction, severe/unstable angina, NYHA class 2 or higher cardiac dysfunction, poorly controlled arrhythmias (including QTcF interval men >450 ms, women >470 ms, QTcF interval calculated by Fridericia formula), symptomatic hyperemia Sexual heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism)
12. High blood pressure, and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90 mmHg)
13. Abnormal coagulation (INR > 1.5 × ULN or activated partial thromboplastin time (APTT) > 1.5 × ULN), with bleeding tendency or receiving thrombolysis or anticoagulant therapy.
14. Hereditary or acquired bleeding and thrombosis trends, such as: hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.
15. Obvious hemoptysis in the first 2 months before the study or daily hemoptysis exceed 2.5ml.
16. Significant clinically bleeding symptoms or clear bleeding tendency within 3 months prior to the study, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood (++) and above, or vasculitis.
17. Artery/ venous thrombosis, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism,etc.
18. Long-term anticoagulant therapy with warfarin or heparin or antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day).
19. Severe infection within 4 weeks prior to first drug administration (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever >38.5℃ during screening period/first drug administration.
20. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
21. Participated in any other drug clinical study within 4 weeks prior to first drug administration , or no more than 5 half-lives from the last study.
22. History of psychotropic substance abuse or drug abuse.
23. Sserious physical or mental illness, laboratory abnormalities, increasing risk of participating in the study, interfere with the results of the study, and patients considered by the investigator to be unfit for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival(RFS) | 72 month
  Duration from surgery to tumor recurrence or death for any reason will be recorded to assess the clinical efficacy of Apatinib Mesylate plus PD-1 antibody SHR-1210 for HCC with high incidence of tumor recurrence after radical resection

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhao, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China